CLINICAL TRIAL: NCT06278415
Title: Pilot Prospective Unblinded Randomized Controlled Study Assessing the Efficacy and Safety of Physiologically Based Cord Clamping Versus Standard Delayed Cord Clamping After Elective Scheduled Cesarean Delivery of Full-term Newborn
Brief Title: Physiologically Based Cord Clamping To Improve Neonatal Outcomes After Elective Cesarean Delivery
Acronym: PhyCord1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Fabiola Children's University Hospital (Other)
Collaborators: The Belgian Kids Fund (Unknown); Fonds IRIS-Recherche (Unknown); Ars Statistica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2021/Neonat/PhyCord 1
Record Dates: First submitted 2024-01-11; First posted 2024-02-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Transient Tachypnea of the Newborn
Keywords: Full-term baby; Scheduled c-section; Neonatal respiratory morbidity; Physiological based-cord clamping
MeSH Terms: conditions — Transient Tachypnea of the Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiological based cord clamping (PBCC) (Experimental): In the intervention group, newborns will receive PBCC. The resuscitation table will place in the operating room as close as possible to the mother's pelvis. After the infant is born, the obstetrician holds the infant. Stabilization will start as soon as the infant is placed on the platform. The nurse places the oximeter sensor on the right wrist and ECG electrodes on the chest of the newborn. Local resuscitation guidelines will be in respect of the NLS-ERC 2021 guidelines. Stabilization of the newborn will be performed while the cord is intact and the cord will be clamped after respiratory stabilization will be achieved, deﬁned as the establishment of regular spontaneous breathing, a HR above 100 bpm SpO 2 above 85% while using supplemental oxygen less than 0,3.
  Interventions: Other: Physiological based cord clamping
- Differed cord clamping (DCC) (Active Comparator): In the control group, newborns will receive standard DCC defined as time based and performed at 60 seconds after birth. Then infants will be transferred to a standard resuscitation table located in a stabilization room next to the operating room. Further treatment and intervention required for cardiopulmonary stabilization will be provided on the standard resuscitation table. Stabilization will start as soon as the infant is placed on the resuscitation table. The nurse will place the oximeter sensor on the right wrist and ECG electrodes on the chest of the newborn. Local resuscitation guidelines will be in respect of the NLS-ERC 2021 guidelines. The time to reach the stabilisation described above (a HR above 100 bpm and SpO 2 above 85% while using supplemental oxygen less than 0,3) is recorded. Then, the infant will be placed on the mother's chest or partner's chest, or alternatively, be prepared and transferred to the transport incubator if further neonatal care is needed.
  Interventions: Other: Differed cord clamping

INTERVENTIONS:
Other: Physiological based cord clamping — see Arm Description
  Arms: Physiological based cord clamping (PBCC)
Other: Differed cord clamping — see Arm Description
  Arms: Differed cord clamping (DCC)

SUMMARY:
Before birth, the baby's lungs are filled with fluid and babies do not use the lungs to breathe, as the oxygen comes from the placenta. As delivery approaches, the lungs begin to absorb the fluid. After vaginal delivery, the umbilical cord is clamped and cut after a delay that allows some of the blood in the umbilical cord and placenta to flow back into the baby. Meanwhile, as the baby breathes for the first time, the lungs fill with air and more fluid is pushed out. However, it does not always work out that way. Some babies need to be delivered via cesarean section, a surgical delivery requiring incisions through the abdominal and uterine walls. After cesarean section, the mother is often unable to hold the baby close right away as a result of her own post-surgical care. Moreover, a baby born by planned cesarean section may have breathing problems because of extra fluid staying in the lungs. Thus, the baby must breathe quicker and harder to get enough oxygen enter into the lungs. Although the baby is usually getting better within one or two days, the treatment requires close monitoring, breathing help, and nutritional help as the baby is too tired to suck and swallow milk. Sometimes, the baby cannot recover well and show greater trouble breathing needing intensive care. This further separates the mother and her baby. A possible mean to help the baby to adapt better after cesarean section while staying close to the mother is to delay cord clamping when efficient breathing is established, either spontaneously or after receiving breathing help at birth. In this study, we intend to test this procedure in term infants born by planned cesarean section and see whether the technique helps the baby to better adapt after birth and to better initiate a deep bond with the mother.

DETAILED DESCRIPTION:
The successful transition from fetal to neonatal life is a major physiological challenge that requires the coordination of lung developmental processes, which culminate with the formation of a diffusible alveolar-capillary barrier, adequate pulmonary vasoreactivity, mature surfactant system, and clearance of lung fluid. During fetal life, gas exchange does not take place in fetal lungs but in the placenta. High pulmonary vascular resistance diverts blood flow to the left atrium through the foramen ovale and to the aorta via the ductus arteriosus. The placental circulation receives 30-50 % of the fetal cardiac output and is the major source of venous return to the fetal heart. Therefore, the umbilical venous return determines the preload for the left ventricle. Shortly before birth and during labor, the lungs undergo important transitional changes. The reabsorption of lung fluid within the airways is initiated during labor by adrenaline-induced activation of sodium channels. Uterine contractions during labor and the onset of inspiration after umbilical cord clamping generate a high transpulmonary pressure gradient leading to additional clearance of fluid from the airways into the surrounding tissue . Following the first breath and lung aeration, oxygen-induced vasodilation leads to a sudden rise in pulmonary blood flow and left atrial pressures, which closes the foramen ovale. Meanwhile, systemic vascular resistance increases above the level of pulmonary vascular resistance after placental removal, which reverses blood flow across the ductus arteriosus and induces ductal closure in response to high oxygen tension.

The route of delivery can impact the success of adaptation to extrauterine life. Over the past 30 years, the rate of cesarean deliveries has increased worldwide. In Belgium, this can be as high as 20% of all deliveries. A subset of cesarean deliveries is scheduled in term infants in the absence of spontaneous labor when vaginal delivery is considered as too risky for maternal and/or child health. The so-called iterative cesarean delivery, which is usually considered as a routine and harmless option, can however alter neonatal health. By contrast with vaginal delivery, infants born at term by iterative cesarean delivery have to adapt despite larger volumes of fluid within airways and interstitial tissue resulting from a limited rise in transpulmonary pressure and adrenaline-induced fluid reabsorption. Subsequently, the retention of lung fluid is responsible for transient tachypnea of the newborn, a respiratory distress that is usually considered as mild, transient, and without sequelae. Moreover, infants born by elective cesarean delivery exhibit a higher risk of positive pressure ventilation resuscitation at birth, admission to the neonatal intensive care unit (NICU), and severe hypoxic respiratory failure requiring mechanical ventilation in the most severe cases. In addition to increased neonatal morbidity, iterative cesarean section can impact mother-infant relationship. After vaginal delivery, immediate skin-to-skin contact during the first minute after birth is the natural process recommended to support mother-infant bonding and promote early onset of breastfeeding. Despite efforts made to start skin-to-skin contact as early as possible after cesarean delivery, immediate contact is practically difficult to implement. In our institution, the infant is usually shortly separated from the mother after umbilical cord clamping to provide first care by a pediatrician before returning on the mother's chest or on the father's chest depending on parental wishes and maternal well-being during the operation. The separation between the mother and her newborn can be further extended in the case of NICU admission for transient tachypnea.

Beside the route of delivery, the timing of umbilical cord clamping can profoundly affect the process of neonatal cardiorespiratory transition. Immediate cord clamping reduces the venous return to the heart, which transiently decreases heartbeats, cardiac output and cerebral blood flow before respiration initiates and pulmonary blood flow increases. Delayed cord clamping for longer than 60 seconds improves the transfusion of blood from the placenta to the newborn. Moreover, it can increase neonatal hemoglobin levels, improve long-term iron stores, and improve neurodevelopmental outcomes. Nevertheless, in both clinical research setting and daily practice, delayed cord clamping lasts rarely more than one minute during cesarean section. More recently, another approach, referred to as physiologically based cord clamping (PBCC), has been proposed to delay cord clamping up to 5 minutes after the onset of ventilation. PBCC allows to start lung aeration while on placental support and, therefore, promotes hemodynamic transition by increasing pulmonary blood flow and maintaining left ventricle preload. This strategy has been demonstrated efficient in preterm lambs and is feasible in very preterm infants, via the use of a purpose-designed resuscitation table that allows delayed cord clamping, maintenance of body temperature, and concomitant respiratory support where necessary. First experience has reported good parental acceptance of the procedure. Because PBCC has not been reported in term infants at risk of respiratory distress after birth, the present project aims to assess whether PBCC in term infants born by elective cesarean section would not be inferior to standard umbilical cord clamping with regards to adaptation to extrauterine life, respiratory morbidity, quality of mother-infant bonding, and maternal safety.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women followed-up in Brugmann University Hospital will be eligible to participate if:

1. Scheduled for cesarean delivery (business days and daily working hours)
2. Singleton pregnancy
3. Cesarean section scheduled at or after 37 weeks gestational age

Exclusion Criteria:

1. Fetal anomalies (congenital malformations, anemia, growth restriction with abnormal Dopplers)
2. Abnormal placentation (placenta previa)
3. Signs of fetal distress necessitating an emergency cesarean section
4. Spontaneous labor before cesarean section
5. Maternal health issue including severe anemia (defined as hemoglobin level < 7 g/dL), preeclampsia, and bleeding disorders
6. Maternal refusal of the use of blood products.
7. General anesthesia for cesarian section
8. Planned cord blood banking
9. Total language barrier without possibility of translation

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-01-21 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Rate of neonatal mortality | within 28 days of delivery
Rate of neonatal resuscitation | within first 10 minutes of life
  Neonatal resuscitation is defined as the use of a T-piece resuscitator for continuous airway positive pressure or intermittent positive pressure (with or without oxygen supplementation).
Rate of neonatal respiratory morbidity | within first 24 hours of life
  Neonatal respiratory morbidity includes transient tachypnea of the newborn, air leak syndrome and respiratory distress syndrome.
Number of admission to the NICU or special care baby unit | within first 72 hours of life

SECONDARY OUTCOMES:
Success of PBCC | within first 10 minutes of life
  Measured by the percentage of neonates in whom the procedure will be achieved without issue, identification of failed PBCC, and duration of stabilization with PBCC (defined as spontaneous breathing heart rate >100 bpm, oxygen saturation by pulse oximetry ≥ 85% with inspired oxygen fraction < 0.3).
Time to first breath/cry | post delivery
  Time in seconds
Changes in physiological variables during neonatal transition | within first 10 minutes of life
  Physiological variables include measurements of preductal oxygen saturation by pulse oximetry (in %) and gases, as well as Apgar scores at 1, 5, and 10 minutes.
Changes in physiological variables during neonatal transition | within first 10 minutes of life
  Physiological variables include measurements of respiratory rate and heart rate (in number per minute)
Changes in physiological variables during neonatal transition | within first 10 minutes of life
  Physiological variables include measurements of body temperature (in degrees Celcius)
Changes in physiological variables during neonatal transition | within first 10 minutes of life
  Physiological variables include measurements of umbilical cord venous hemoglobin (in gr/dl)
Changes in physiological variables during neonatal transition | within first 10 minutes of life
  Physiological variables include measurements of umbilical cord pH
Changes in physiological variables during neonatal transition | within first 10 minutes of life
  Physiological variables include measurements of Apgar scores (from 1 to 10 units on the scale, the highest scores meaning better outcome) at 1, 5 and 10 minutes
Early neonatal parameters | within the first 3 hours of life
  Early neonatal parameters include body temperature (in degrees Celcius) at 1, 2 and 3 hours of life.
Early neonatal parameters | within first 24 hours of life
  Early neonatal parameters include body weight (in gramme).
Hemoglobin level | at 48 hours of life
  in g/dl
Bilirubin level | at 48 hours of life
  in mg/dl
Number of neonatal adverse events | within first 72 hours of live
  including hypoglycemia, sepsis, and the need for phototherapy.
Maternal perioperative parameters | at Day 1 post delivery
  Maternal perioperative parameters include total surgical time (in minutes), intraoperative intravenous fluid volume, intraoperative blood loss, uterotonic administration, and postoperative hemoglobin level at day 1.
Maternal perioperative parameters | at Day 1 post delivery
  Maternal perioperative parameters include intraoperative intravenous fluid volume and intraoperative blood loss (in ml), uterotonic administration, and postoperative hemoglobin level at day 1.
Maternal perioperative parameters | at Day 1 post delivery
  Maternal perioperative parameters include uterotonic administration (Yes/No), and postoperative hemoglobin level at day 1.
Maternal perioperative parameters | at Day 1 post delivery
  Maternal perioperative parameters include postoperative hemoglobin level (in gr/dl).
Number of maternal adverse events | within first 2 weeks post delivery
  Maternal adverse events include death, blood transfusion, postpartum hemorrhage, hysterectomy, admission in the Intensive Care Unit, wound seroma, and wound cellulitis.
Rate of maternal-infant bonding | up to 2 weeks post delivery
  breastfeeding (yes/no)
Rate of maternal-infant bonding | at 2 weeks post delivery
  maternal depression (measured by the Edinburgh Postnatal Depression Scale (EPDS) - score min = 0, score max = 30, higher score = worse outcome)
Rate of maternal-infant bonding | at 2 weeks post delivery
  maternal depression (measured by the Maternal Infant Bonding Scale (MIBS) - score min = 0, score max = 24, higher score = worse outcome)
Child developmental assessment | at 2 weeks postnatally
  The child developmental assessment is done using the Brazelton Neonatal Behavioral Assessment Scale (NBAS) - score min = 1, score max = 6, higher score = better outcome
Parental satisfaction survey | at 2 weeks post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Anna AMORUSO, Principal Investigator — HUDERF
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - Hôpital Universitair Des Enfants Reine Fabiola, Brussels